CLINICAL TRIAL: NCT02101268
Title: A Phase 3, Randomized Study To Evaluate the Efficacy of Momelotinib Versus Best Available Therapy in Anemic or Thrombocytopenic Subjects With Primary Myelofibrosis, Post-polycythemia Vera Myelofibrosis, or Post-essential Thrombocythemia Myelofibrosis Who Were Treated With Ruxolitinib
Brief Title: Efficacy of Momelotinib Versus Best Available Therapy in Anemic or Thrombocytopenic Subjects With Primary Myelofibrosis (MF), Post-polycythemia Vera MF, or Post-essential Thrombocythemia MF
Acronym: Simplify 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-352-1214; 2013-005007-13 (EudraCT Number)
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Results first posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Primary Myelofibrosis (PMF); Post-polycythemia Vera (Post-PV); Post-essential Thrombocythemia Myelofibrosis (Post-ET MF)
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Momelotinib (Experimental): Participants will receive open-label momelotinib for 24 weeks during the randomized treatment phase, after which they will be eligible to receive momelotinib in an extended treatment phase for up to an additional 204 weeks.
  Interventions: Drug: Momelotinib
- Arm 2: Best Available Therapy (BAT) (Active Comparator): Participants in the BAT treatment arm will receive open-label treatment at doses and schedules determined by the investigator in accordance with standard of care. Therapy may be changed at any time during the study except during the screening period. After completion of the randomized treatment phase, participants will be eligible to receive momelotinib for the duration of the study during the extended treatment phase for up to 204 weeks.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: Momelotinib — Momelotinib tablet administered orally once daily
  Other Names: GS-0387; CYT387
  Arms: Arm 1: Momelotinib
Drug: Best Available Therapy (BAT) — Regimens for BAT may include but are not limited to chemotherapy (eg hydroxyurea), anagrelide, corticosteroid, hematopoietic growth factor, immunomodulating agent, androgen, interferon, and may include no myelofibrosis treatment.
  Arms: Arm 2: Best Available Therapy (BAT)

SUMMARY:
This study is to determine the efficacy of momelotinib (MMB) versus best available therapy (BAT) in anemic or thrombocytopenic adults with primary myelofibrosis (PMF), or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (Post-PV/ET MF) who were treated with ruxolitinib as measured by splenic response rate at Week 24 (SRR24).

Participants will be randomized to receive either MMB or BAT for 24 weeks during the randomized treatment phase, after which they will be eligible to receive MMB in an extended treatment phase for up to an additional 204 weeks. After discontinuation of study medication, assessments will continue for 12 additional weeks, after which participants will be contacted for survival follow-up approximately every 6 months for up to 5 years from the date of enrollment or until study termination. For those subjects planning to continue treatment with MMB following the end of the study, the End of Treatment, 30-day, 12-Week, and survival follow-up visits are not required.

ELIGIBILITY:
Key Inclusion Criteria:

* Palpable splenomegaly at least 5 cm below left costal margin
* Confirmed diagnosis of PMF in accordance, or Post-PV/ET MF
* Currently or previously treated with ruxolitinib for PMF or Post-PV/ET MF for at least 28 days, and characterized by

  * Requirement for RBC transfusion while on ruxolitinib treatment, OR
  * Dose adjustment of ruxolitinib to < 20 mg twice daily at start of or during ruxolitinib treatment AND at least one of the following while on ruxolitinib treatment:

    * ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 thrombocytopenia, OR
    * ≥ CTCAE Grade 3 anemia, OR
    * ≥ CTCAE Grade 3 hematoma (bleed)
* High risk OR intermediate-2 risk as defined by Dynamic International Prognostic Scoring System (DIPSS), OR intermediate-1 risk as defined by DIPSS and associated with symptomatic splenomegaly, and/or hepatomegaly
* If receiving myelofibrosis therapy, must be on a stable dose of the same regimen for at least 2 weeks prior to screen date and through the screening period
* If not receiving myelofibrosis therapy, must remain off therapy for at least 2 weeks prior to screen date and through the screening period
* Acceptable laboratory assessments obtained within 14 days prior to Randomization

  * Absolute neutrophil count (ANC) > 0.75 x 10^9/L in the absence of growth factor in the prior 7 days
  * Peripheral blood blast count < 10%
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x the upper limit of the normal range (ULN) (≤ 5 x ULN if liver is involved by extramedullary hematopoiesis as judged by the investigator or if related to iron chelator therapy that was started within the prior 60 days)
  * Calculated creatinine clearance of ≥ 45 mL/min
  * Direct bilirubin ≤ 2.0 x ULN
* Life expectancy > 24 weeks
* Negative serum pregnancy test for female subjects (unless surgically sterile or greater than two years post-menopausal)
* Males and females of childbearing potential must agree to use protocol-specified method(s) of contraception
* Females who are nursing must agree to discontinue nursing before the first dose of MMB
* Able to understand and willing to sign informed consent form (ICF)

Key Exclusion Criteria:

* Prior splenectomy
* Splenic irradiation within 3 months prior to Randomization
* Use of investigational agent within 28 days prior to Randomization
* Prior treatment with MMB
* Hematopoietic growth factor (granulocyte growth factor, erythropoiesis stimulating agent, thrombopoietin mimetic) within 28 days prior to Randomization
* Uncontrolled inter-current illness, per protocol
* Known positive status for human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier
* Presence of peripheral neuropathy ≥ CTCAE Grade 2
* Unwilling or unable to undergo a MRI or CT Scan per study protocol requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-06-19 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (48):
- United States (13):
  - Los Angeles, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Kansas City, Kansas
  - Baltimore, Maryland
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Houston, Texas
- Canada (3):
  - Edmonton, Alberta
  - Montreal
  - Toronto
- France (7):
  - Lille
  - Marseille
  - Nantes
  - Paris
  - Pierre-Bénite
  - Toulouse
  - Villejuif
- Germany (4):
  - Cologne
  - Dresden
  - Hamburg
  - Mannheim
- Israel (4):
  - Ashkelon
  - Haifa
  - Jerusalem
  - Tel Aviv
- Italy (7):
  - Bologna
  - Florence
  - Genova
  - Milan
  - Novara
  - Roma
  - Varese
- Spain (6):
  - Badalona
  - Barcelona
  - Madrid
  - Salamanca
  - Valencia
  - Zaragoza
- United Kingdom (4):
  - Birmingham, England
  - Leeds, England
  - Leicester, England
  - London, England

REFERENCES:
- [Derived] Mesa RA, Talpaz M, Mazerolle F, Gorsh B, M'Hari M, Regnault A, Ellis C, Wang Z, Purser M, Liu T, Strouse B, Patnaik D. Time Without Transfusion Reliance (TWiTR): Integrating Survival Quality Into Myelofibrosis Treatment Strategies Based on the Phase 3 SIMPLIFY-1, SIMPLIFY-2, and MOMENTUM Trials. EJHaem. 2025 Jun 18;6(3):e70075. doi: 10.1002/jha2.70075. eCollection 2025 Jun. PMID 40535755
- [Derived] Harrison CN, Mesa R, Talpaz M, Gupta V, Gerds AT, Perkins A, Goh YT, Fox ML, McLornan D, Palmer J, Foltz L, Vannucchi A, Koschmieder S, Passamonti F, Lee SE, Ellis C, Strouse B, Gonzalez Carreras FJ, Oh ST. Longitudinal Assessment of Transfusion Intensity in Patients With JAK Inhibitor-Naive or -Experienced Myelofibrosis Treated With Momelotinib. Clin Lymphoma Myeloma Leuk. 2025 Mar;25(3):199-211. doi: 10.1016/j.clml.2024.10.001. Epub 2024 Oct 16. PMID 39516087
- [Derived] Harrison CN, Vannucchi AM, Recher C, Passamonti F, Gerds AT, Hernandez-Boluda JC, Yacoub A, Sirhan S, Ellis C, Patel B, Strouse B, Platzbecker U. Momelotinib versus Continued Ruxolitinib or Best Available Therapy in JAK Inhibitor-Experienced Patients with Myelofibrosis and Anemia: Subgroup Analysis of SIMPLIFY-2. Adv Ther. 2024 Sep;41(9):3722-3735. doi: 10.1007/s12325-024-02928-4. Epub 2024 Jul 11. PMID 38990433
- [Derived] Verstovsek S, Mesa R, Gupta V, Lavie D, Dubruille V, Cambier N, Platzbecker U, Hus M, Xicoy B, Oh ST, Kiladjian JJ, Vannucchi AM, Gerds A, Egyed M, Mayer J, Sacha T, Kawashima J, Morris M, Huang M, Harrison C. Momelotinib long-term safety and survival in myelofibrosis: integrated analysis of phase 3 randomized controlled trials. Blood Adv. 2023 Jul 25;7(14):3582-3591. doi: 10.1182/bloodadvances.2022009311. PMID 37042865
- [Derived] Harrison CN, Vannucchi AM, Platzbecker U, Cervantes F, Gupta V, Lavie D, Passamonti F, Winton EF, Dong H, Kawashima J, Maltzman JD, Kiladjian JJ, Verstovsek S. Momelotinib versus best available therapy in patients with myelofibrosis previously treated with ruxolitinib (SIMPLIFY 2): a randomised, open-label, phase 3 trial. Lancet Haematol. 2018 Feb;5(2):e73-e81. doi: 10.1016/S2352-3026(17)30237-5. Epub 2017 Dec 20. PMID 29275119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 156 participants were randomized at 52 centers in 8 countries.
Pre-assignment Details: Participants were screened within 30 days before randomization to determine eligibility for participation in the study. Participants who were not randomized within the 30-day screening window were considered screen failures. At randomization, participants were randomly assigned 2:1 to MMB:BAT.
Groups:
- Momelotinib (MMB): Participants received momelotinib orally once daily at a starting dose of 200 mg. Additional available strengths included 100 mg and 150 mg.
- Best Available Therapy (BAT): Participants received treatment at doses and schedules determined by the investigator in accordance with standard of care. Therapy may have been changed at any time during the study except during the screening period. No active therapy was a permissible option.
- MMB to MMB: After completion of the 24-week randomized treatment phase, participants randomized to the MMB group who tolerated and derived clinical benefit from MMB had the option to receive MMB at their current dose in an extended treatment phase for up to an additional 204 weeks. Available strengths included 100 mg, 150 mg and 200 mg.
- BAT to MMB: After completion of the 24-week randomized treatment phase, participants randomized to the BAT treatment arm had the option to receive MMB 200 mg once daily in an extended treatment phase for up to an additional 204 weeks. Additional available strengths included 100 mg and 150 mg.
Period: Randomized Treatment Phase
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT) | MMB to MMB | BAT to MMB
Started | 104 (The MMB group is only applicable to the randomized treatment phase. Participants who complete the randomized phase and continue to receive MMB in the extended treatment phase constitute the MMB to MMB group.) | 52 (The BAT group is only applicable to the randomized treatment phase. Participants who complete the randomized phase and begin receiving MMB in the extended treatment phase constitute the BAT to MMB group.) | 0 (The MMB to MMB group is only applicable to the extended treatment phase.) | 0 (The BAT to MMB group is only applicable to the extended treatment phase.)
Completed | 77 | 41 | 0 | 0
Not Completed | 27 | 11 | 0 | 0
Not completed — Subject Decision | 8 | 4 | 0 | 0
Not completed — Physician Decision | 4 | 1 | 0 | 0
Not completed — Symptomatic Spleen Growth | 0 | 1 | 0 | 0
Not completed — Adverse Event | 6 | 0 | 0 | 0
Not completed — Death | 5 | 4 | 0 | 0
Not completed — Disease Progression | 4 | 1 | 0 | 0
Period: Extended Treatment Phase
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT) | MMB to MMB | BAT to MMB
Started | 0 (The MMB group is only applicable to the randomized treatment phase. Participants who complete the randomized phase and continue to receive MMB in the extended treatment phase constitute the MMB to MMB group.) | 0 (The BAT group is only applicable to the randomized treatment phase. Participants who complete the randomized phase and begin receiving MMB in the extended treatment phase constitute the BAT to MMB group.) | 64 (Of 77 participants in the MMB group who completed the randomized treatment phase, 64 entered the extended treatment phase to continue receiving MMB.) | 40 (Of 41 participants in the BAT group who completed the randomized treatment phase, 40 entered the extended treatment phase to begin receiving MMB.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 64 | 40
Not completed — Subject Decision | 0 | 0 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 14 | 18
Not completed — Death | 0 | 0 | 5 | 1
Not completed — Transferred to Study SRA-MMB-4365 | 0 | 0 | 15 | 7
Not completed — Disease Progression | 0 | 0 | 13 | 6
Not completed — Lack of Efficacy | 0 | 0 | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 104 | 52 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 14 | 55
  >=65 years | 63 | 38 | 101
Age, Continuous [Median (Full Range); unit: years] | 67.0 [41 to 92] | 69.5 [52 to 82] | 68.0 [41 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 69 | 24 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 81 | 40 | 121
  Unknown or Not Reported | 18 | 8 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 83 | 44 | 127
  Black or African American | 6 | 0 | 6
  Not Permitted | 15 | 8 | 23
Transfusion Dependent [Count of Participants; unit: Participants]
  Yes | 58 | 27 | 85
  No | 46 | 25 | 71
Total Symptom Score (TSS) [Count of Participants; unit: Participants] — See secondary outcome description
  Participants
    < 18 | 61 | 28 | 89
    >= 18 | 43 | 24 | 67
Weight [Median (Inter-Quartile Range); unit: kg] | 75.4 [68.0 to 87.0] | 74.0 [62.0 to 81.3] | 75.0 [66.0 to 85.7]
Height [Median (Inter-Quartile Range); unit: cm] | 170.0 [164.0 to 177.8] | 168.0 [160.0 to 175.0] | 170.0 [162.5 to 176.0]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 25.9 [23.6 to 28.2] | 26.1 [23.5 to 29.1] | 26.0 [23.6 to 28.6]
Hemoglobin [Median (Inter-Quartile Range); unit: g/dL] | 9.0 [7.9 to 10.7] | 9.2 [8.5 to 10.1] | 9.0 [8.1 to 10.6]

OUTCOME MEASURES:

1. Primary Outcome: Splenic Response Rate at Week 24
Description: Splenic response rate at Week 24 is defined as the percentage of participants who achieved a spleen volume reduction of ≥ 35% from baseline at the Week 24 assessment as measured by MRI or CT.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT)
Number analyzed (Participants) | 104 | 52
Participants
  Responder | 7 | 3
  Nonresponder | 97 | 49
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.90, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.01, 95% CI 2-sided [-0.09 to 0.10]

2. Secondary Outcome: Total Symptom Score (TSS) Response Rate at Week 24
Description: Total symptom score (TSS) is defined as the percentage of participants who achieved a ≥50% reduction in TSS at Week 24 versus baseline as measured by the modified Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) v2.0 diary. Response rate was calculated using the average of the daily TSS from a consecutive 28-day period prior to Week 24, which had ≥20 daily TSS available.
  The modified MPN-SAF patient-reported outcome instrument consisted of 8 items assessing worst daily incidence of tiredness, filling up quickly, abdominal discomfort, night sweats, itching, bone pain, pain under ribs on left side, and inactivity. Scoring of TSS in this study was based on 7 of these items, (0-70) excluding inactivity. These items assess the impact experienced by the participant in the 24 hours prior to completing the questionnaire. All items are measured using a 0 to 10 Numeric Rating Scale, with 0 corresponding to "Absent" and 10 corresponding to "Worst Imaginable."
Time Frame: Week 24
Population: TSS rate analysis at Week 24 only included participants with TSS > 0 at baseline or with TSS = 0 at baseline but with TSS > 0 or missing at Week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT)
Number analyzed (Participants) | 103 | 51
Participants
  Responder | 27 | 3
  Nonresponder | 76 | 48
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Best Available Therapy (BAT); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.20, 95% CI 2-sided [0.09 to 0.32]

3. Secondary Outcome: Rate of Red Blood Cell (RBC) Transfusion in the Randomized Treatment Phase, (the Average Number of RBC Units Transfused Per Month Not Associated With Overt Bleeding)
Description: Rate of RBC transfusion is defined as the average number of RBC units transfused not associated with clinically overt bleeding per subject-month during the randomized treatment Phase.
Time Frame: Baseline to Week 24
Measure: Median (Inter-Quartile Range); unit: units/month
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT)
Number analyzed (Participants) | 104 | 52
units/month | 0.5 [0.0 to 2.4] | 1.2 [0.0 to 2.8]
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.38, Negative Binomial Model, Adjusted; Rate ratio = 0.80, 95% CI 2-sided [0.49 to 1.31] — A smaller ratio represents larger benefit

4. Secondary Outcome: RBC Transfusion Independence Rate at Week 24, (Defined as Absence of RBC Transfusions and no Hemoglobin Level Below 8 g/dL in the 12 Weeks Prior to Week 24, Excluding Cases Associated With Clinically Overt Bleeding)
Description: RBC transfusion independence rate is the percentage of participants who achieved transfusion independence at Week 24 (responders). RBC transfusion independence is defined as absence of RBC transfusions and no hemoglobin level below 8 g/dL in the 12 weeks prior to Week 24, excluding cases associated with clinically overt bleeding. Transfusion dependence, (non-responder) is defined as at least 4 units of RBC transfusion, or a Hgb level below 8 g/dL, in the 8 weeks prior to week 24.
  Methods used to assess this outcome measure include collection and recording of any instances of RBC transfusions and collection and recording of any local or central lab hemoglobin measurements
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT)
Number analyzed (Participants) | 104 | 52
Participants
  Responder | 45 | 11
  Nonresponder | 59 | 41
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = 0.23, 95% CI 2-sided [0.09 to 0.37] — A larger proportion represents larger benefit

5. Secondary Outcome: RBC Transfusion Dependence Rate at Week 24
Description: RBC transfusion dependence is the percentage of participants who are transfusion dependent at Week 24, defined as at least 4 units of RBC transfusions, or a hemoglobin level below 8 g/dL in the 8 weeks prior to Week 24, excluding cases associated with clinically overt bleeding.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT)
Number analyzed (Participants) | 104 | 52
Participants
  Dependent | 52 | 33
  Nondependent | 52 | 19
Statistical Analysis 1: Comparison: Momelotinib (MMB) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.10, Cochran-Mantel-Haenszel; Proportion Difference - Stratified CMH = -0.13, 95% CI 2-sided [-0.29 to 0.03] — A smaller proportion represents larger benefit

ADVERSE EVENTS:
Time Frame: Serious and other Adverse events were recorded that occurred from initiation of investigational product (IP) until 30 days after the last administration of IP regardless of cause or relationship. Serious events are monitored up to 12 weeks and all-cause mortality was assessed for up to 5 years.
Arm/Group | Momelotinib (MMB) | Best Available Therapy (BAT) | MMB to MMB | BAT to MMB
All-Cause Mortality (participants affected / at risk) | 8/104 | 5/52 | 29/64 | 18/40
Serious Adverse Events (participants affected / at risk) | 37/104 | 12/52 | 33/64 | 19/40
Other Adverse Events (participants affected / at risk) | 99/104 | 46/52 | 63/64 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=104) | Best Available Therapy (BAT) (N=52) | MMB to MMB (N=64) | BAT to MMB (N=40)
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 6 | 1
Sepsis (Infections and infestations) | 2 | 2 | 4 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 1 | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Visceral venous thrombosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 1 | 4
Spontaneous haematoma (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
General physical health deterioration (General disorders) | 2 | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 2 | 3
Generalised oedema (General disorders) | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Momelotinib (MMB) (N=104) | Best Available Therapy (BAT) (N=52) | MMB to MMB (N=64) | BAT to MMB (N=40)
Diarrhoea (Gastrointestinal disorders) | 33 | 8 | 19 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 6 | 17 | 8
Asthenia (General disorders) | 20 | 11 | 8 | 11
Pyrexia (General disorders) | 13 | 4 | 16 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 6 | 8 | 11
Nausea (Gastrointestinal disorders) | 20 | 5 | 8 | 5
Anaemia (Blood and lymphatic system disorders) | 15 | 10 | 14 | 6
Fatigue (General disorders) | 16 | 10 | 7 | 7
Abdominal pain (Gastrointestinal disorders) | 16 | 7 | 7 | 5
Oedema peripheral (General disorders) | 11 | 6 | 10 | 6
Dizziness (Nervous system disorders) | 16 | 4 | 6 | 6
Headache (Nervous system disorders) | 16 | 3 | 4 | 6
Urinary tract infection (Infections and infestations) | 11 | 4 | 8 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 5 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 3 | 8 | 5
Weight decreased (Investigations) | 10 | 3 | 7 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 0 | 6 | 7
Constipation (Gastrointestinal disorders) | 11 | 2 | 5 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 8 | 4 | 3 | 6
Decreased appetite (Metabolism and nutrition disorders) | 7 | 2 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 4 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 3
Bronchitis (Infections and infestations) | 5 | 2 | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 1 | 5 | 2
Hypertension (Vascular disorders) | 10 | 2 | 5 | 2
Paraesthesia (Nervous system disorders) | 8 | 1 | 4 | 3
Vomiting (Gastrointestinal disorders) | 7 | 1 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1 | 2 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 2 | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 7 | 1
Dyspepsia (Gastrointestinal disorders) | 10 | 1 | 2 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 7 | 2 | 6 | 1
Blood creatinine increased (Investigations) | 6 | 0 | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 1 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 5 | 3 | 2
Insomnia (Psychiatric disorders) | 3 | 4 | 4 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 2
Contusion (Injury, poisoning and procedural complications) | 5 | 3 | 2 | 2
Hypotension (Vascular disorders) | 3 | 2 | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 5 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3 | 2
Oral herpes (Infections and infestations) | 7 | 0 | 2 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 1 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2 | 2 | 3
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 3
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 1
Ascites (Gastrointestinal disorders) | 4 | 2 | 2 | 2
Early satiety (General disorders) | 3 | 6 | 2 | 1
Haematoma (Vascular disorders) | 0 | 0 | 2 | 4
Chills (General disorders) | 2 | 0 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 2 | 2
Melaena (Gastrointestinal disorders) | 1 | 1 | 2 | 2
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 3
Cardiac failure (Cardiac disorders) | 1 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 2
Splenomegaly (Blood and lymphatic system disorders) | 2 | 3 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Best available therapy could also include the approved JAK inhibitor, ruxolitinib, and 88% of participants in the BAT arm continued to receive ruxolitinib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements varied with individual investigators, but did not prohibit any investigator from publishing. Investigators were not to publish results of the study until a period of time (eg. 2 years) following completion of the trial at all participating institutions but could do so earlier with consent of the Sponsor.